CLINICAL TRIAL: NCT02853864
Title: Influence of Gender on Interaction of Propofol and Dexmedetomidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Intravenous anesthesia
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2016-12

CONDITIONS: Anesthesia
Keywords: Gender; Propofol; Dexmedetomidine; Interaction
MeSH Terms: conditions — Coitus | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Propofol and 0.0 ng/ml Dexmedetomidine (Placebo Comparator): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.0ng/ml administered for 15min, and increased by 0.2 ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.0 ng/ml Dexmedetomidine; Drug: Propofol
- Propofol and 0.4 ng/ml Dexmedetomidine (Experimental): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.4ng/ml administered for 15min, and increased by 0.2 ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.4 ng/ml Dexmedetomidine; Drug: Propofol
- Propofol and 0.6 ng/ml Dexmedetomidine (Experimental): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.6ng/ml administered for 15min, and increased by 0.2 ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.6 ng/ml Dexmedetomidine; Drug: Propofol
- Propofol and 0.8 ng/ml Dexmedetomidine (Experimental): Propofol infusion was started to provide an effect-site concentration of 1.0ug/ml after Dexmedetomidine which target plasma concentration is 0.8ng/ml administered for 15min, and increased by 0.2 ug/ml until the patient's consciousness disappears.
  Interventions: Drug: 0.8 ng/ml Dexmedetomidine; Drug: Propofol

INTERVENTIONS:
Drug: 0.0 ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.0 ng/ml
  Arms: Propofol and 0.0 ng/ml Dexmedetomidine
Drug: 0.4 ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.4 ng/ml
  Arms: Propofol and 0.4 ng/ml Dexmedetomidine
Drug: 0.6 ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.6 ng/ml
  Arms: Propofol and 0.6 ng/ml Dexmedetomidine
Drug: 0.8 ng/ml Dexmedetomidine — Dexmedetomidine target plasma concentration is 0.8 ng/ml
  Arms: Propofol and 0.8 ng/ml Dexmedetomidine
Drug: Propofol — The propofol infusion was started to provide an effect-site concentration of 1.0 ug/ml, and increased by 0.2 ug/ml until loss of consciousness

SUMMARY:
The purpose of this study is to determine the effect of gender on pharmacodynamic interaction of propofol and dexmedetomidine, exploring the effect of gender on propofol unconsciousness median effective concentration with different dose dexmedetomidine.

DETAILED DESCRIPTION:
60 cases male patients were randomly divided into four groups,and 60 female patients were also randomly divided into four groups.In each group, dexmedetomidine target plasma concentration are 0,0.4,0.6,0.8 ng/ml. Dexmedetomidine administered 15 min before target controlled infusion of propofol. The propofol infusion is started to provide a target effect-site concentration of 1.0 ug/ml, and increased by 0.2 ug/ml until loss of consciousness when the effect-site concentration and target concentration are equilibrium.

ELIGIBILITY:
Inclusion Criteria:

1. Weight:18≦ BMI≦25
2. Written informed consent from the patient or the relatives of the participating patient.

Exclusion Criteria:

1. A previous history of intolerance to the study drug or related compounds and additives.
2. Existing significant haematological, endocrine, metabolic or gastrointestinal disease.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
the effect-site EC50 of propofol on loss of consciousness with different gender | within 30 min during the induction of anesthesia
  The aim of the investigators study is to define the optimum target concentration (EC50) of propofol for loss of consciousness with different dexmedetomidine target plasm concentration.

SECONDARY OUTCOMES:
The EC95 of propofol for loss of consciousness with different gender | within 30 min during the induction of anesthesia
  The aim of the investigators study is to define the optimum target concentration (EC95) of propofol for loss of consciousness with different dexmedetomidine target plasm concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodaka M, Johansen JW, Sebel PS. The influence of gender on loss of consciousness with sevoflurane or propofol. Anesth Analg. 2005 Aug;101(2):377-381. doi: 10.1213/01.ANE.0000154534.71371.4F. PMID 16037147